CLINICAL TRIAL: NCT02406209
Title: A Phase 2 Randomized, Investigator-Masked, Comparator-controlled Trial to Evaluate the Safety and Efficacy of NS2 Eye Drops in Patients With Anterior Uveitis
Brief Title: A Safety and Efficacy Study of NS2 in Patients With Anterior Uveitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NS2-02
Record Dates: First submitted 2015-03-26; First posted 2015-04-02 (Estimated); Results first posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2019-02

CONDITIONS: Non-infectious Anterior Uveitis
Keywords: uveitis; acute uveitis; anterior uveitis; NS2; Aldeyra; prednisolone acetate
MeSH Terms: conditions — Uveitis; Uveitis, Anterior | interventions — prednisolone acetate

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- NS2 (Experimental): NS2 ophthalmic drops (0.5%) in the affected eye
  Interventions: Drug: NS2
- NS2 and Pred Forte (Experimental): NS2 ophthalmic drops (0.5%) and Prednisolone acetate ophthalmic suspension (1%) in the affected eye
  Interventions: Drug: NS2; Drug: Prednisolone acetate ophthalmic suspension (1%)
- Pred Forte (Active Comparator): Prednisolone acetate ophthalmic suspension (1%) in the affected eye
  Interventions: Drug: Prednisolone acetate ophthalmic suspension (1%)

INTERVENTIONS:
Drug: NS2 — NS2 ophthalmic drops (0.5%)
  Arms: NS2; NS2 and Pred Forte
Drug: Prednisolone acetate ophthalmic suspension (1%)
  Other Names: Pred Forte
  Arms: NS2 and Pred Forte; Pred Forte

SUMMARY:
This is a randomized, multi-center, investigator masked, comparator controlled study. The purpose of this study is to determine the efficacy and safety of NS2 in patients with non-infectious acute anterior uveitis. Subjects will be randomized 1:1:1 to receive multiple doses of NS2 0.5%, NS2 0.5% and Pred Forte® 1%, or Pred Forte® 1%.

Free aldehydes are thought to be related to inflammatory diseases such as uveitis. NS2, a small molecule aldehyde trap, may decrease inflammation by lowering aldehyde levels.

ELIGIBILITY:
Inclusion Criteria:

* Non-infectious anterior uveitis
* Grade 1 - Grade 3 anterior chamber cell count
* Subjects must have Intraocular pressure <25 mmHg at baseline and may only administer a maximum of 1 topical medication to control Intraocular pressure in the study eye.
* Visual acuity ≥ 20/200 in the study eye

Exclusion Criteria:

* Severe/serious ocular pathology
* Active intermediate or posterior uveitis.
* Previous anterior uveitis episode in the study eye within 4 weeks of Visit 1
* Oral corticosteroids within 14 days of Visit 1
* Intravitreal or sub-Tenon corticosteroid treatment in the study eye within the past 6 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C.Stephen Foster, MD, FACS, FACR, Principal Investigator — Massachusetts Eye Research and Surgery Institution
Locations (15):
- United States (15):
  - Hull Eye Center, Lancaster, California
  - Colorado Retina Associates,PC, Golden, Colorado
  - Eye Center of Southern Connecticut, Hamden, Connecticut
  - Bascom Palmer Eye Institute, Plantation, Florida
  - Valley Eye Physicians & Surgeons, Ayer, Massachusetts
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Massachusetts Eye Research and Surgery Institution (MERSI), Waltham, Massachusetts
  - Oakland Ophthalmic Surgery, Birmingham, Michigan
  - Lifelong Vision Foundation, Chesterfield, Missouri
  - Tauber Eye Center, Kansas City, Missouri
  - UNMC Stanley Truhlsen Eye Institute, Omaha, Nebraska
  - Metropolitan Eye Research & Surgery Institute, Palisades Park, New Jersey
  - Mid-Atlantic Retina, Philadelphia, Pennsylvania
  - Houston Eye Associates, Houston, Texas
  - Virginia Eye Consultants, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mandell KJ, Clark D, Chu DS, Foster CS, Sheppard J, Brady TC. Randomized Phase 2 Trial of Reproxalap, a Novel Reactive Aldehyde Species Inhibitor, in Patients with Noninfectious Anterior Uveitis: Model for Corticosteroid Replacement. J Ocul Pharmacol Ther. 2020 Dec;36(10):732-739. doi: 10.1089/jop.2020.0056. Epub 2020 Sep 22. PMID 32955967

RESULTS

PARTICIPANT FLOW:
Groups:
- NS2 Ophthalmic Drops (0.5%): NS2 administered four times daily (QID) for approximately 6 weeks
- NS2 (0.5%) and Pred Forte® (0.1%) Ophthalmic Drops: NS2 QID for approximately 6 weeks and Pred Forte® twice daily (BID) tapered through Week 4
- Pred Forte® (1%) Ophthalmic Drops: Pred Forte® QID tapered through Week 6
Period: Overall Study
Arm/Group | NS2 Ophthalmic Drops (0.5%) | NS2 (0.5%) and Pred Forte® (0.1%) Ophthalmic Drops | Pred Forte® (1%) Ophthalmic Drops
Started | 15 | 16 | 14
Completed | 7 | 7 | 6
Not Completed | 8 | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NS2 Ophthalmic Drops (0.5%) | NS2 (0.5%) and Pred Forte® (0.1%) Ophthalmic Drops | Pred Forte® (1%) Ophthalmic Drops | Total
Number analyzed (Participants) | 15 | 16 | 14 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (13.84) | 48.0 (19.49) | 40.9 (11.38) | 45.4 (15.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 8 | 32
  Male | 5 | 2 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 2 | 11
  White | 8 | 12 | 12 | 32
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 3
  Not Hispanic or Latino | 12 | 16 | 14 | 42
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 16 | 14 | 45
Height [Mean (Standard Deviation); unit: centimeters] | 168.9 (14.45) | 165.7 (9.38) | 168.6 (10.24) | 167.7 (11.39)
Weight [Mean (Standard Deviation); unit: kilograms] | 79.7 (18.53) | 78.5 (25.04) | 78.3 (22.46) | 78.8 (21.74)

OUTCOME MEASURES:

1. Primary Outcome: Anterior Chamber Cell Grade at Week 8
Description: Change from baseline comparison of NS2 ophthalmic drops (0.5%), NS2 (0.5%) and Pred Forte® (0.1%) ophthalmic drops, and Pred Forte® (1%) ophthalmic drops on an anterior chamber cell grade scale of 0 to 4 (0 = absent, 4 = severe). The least squares mean (standard error) was derived from analysis of covariance (ANCOVA) with baseline as a covariate and treatment group as a factor.
Time Frame: The efficacy assessment period was assessed at Week 8; baseline was Day 1.
Population: Modified intent-to-treat
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NS2 Ophthalmic Drops (0.5%) | NS2 (0.5%) and Pred Forte® (0.1%) Ophthalmic Drops | Pred Forte® (1%) Ophthalmic Drops
Number analyzed (Participants) | 15 | 16 | 13
units on a scale | -0.7 (0.31) | -0.9 (0.29) | -0.5 (0.32)

ADVERSE EVENTS:
Time Frame: The period of time over which adverse events were collected for each subject in the clinical trial was approximately nine weeks.
Arm/Group | NS2 Ophthalmic Drops (0.5%) | NS2 (0.5%) and Pred Forte® (0.1%) Ophthalmic Drops | Pred Forte® (1%) Ophthalmic Drops
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 8/15 | 8/16 | 3/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NS2 Ophthalmic Drops (0.5%) (N=15) | NS2 (0.5%) and Pred Forte® (0.1%) Ophthalmic Drops (N=16) | Pred Forte® (1%) Ophthalmic Drops (N=14)
Iridocyclitis (Eye disorders) | 0 | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0
Cystoid macular oedema (Eye disorders) | 0 | 1 | 0
Eye inflammation (Eye disorders) | 0 | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0
Macular oedema (Eye disorders) | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Head discomfort (Nervous system disorders) | 1 | 0 | 0
Photophobia (Nervous system disorders) | 1 | 0 | 0
Visual acuity reduced (Nervous system disorders) | 1 | 0 | 0
Ligament rupture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Ligament sprain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Syncope (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
General disorders and administration site conditions (General disorders) | 6 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes